CLINICAL TRIAL: NCT05572853
Title: Analysis of Electrical Activity of Respiratory Muscles in Patients Undergoing Oxygen Therapy With COVID-19: Cross-sectional Study
Brief Title: Respiratory Muscles Electromyography in Patients With Covid-19
Acronym: EMG-COVID
Status: Completed | Type: Observational
Sponsor: University of Pernambuco (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Shirley Lima Campos, Associate Professor, University of Pernambuco
Other Study IDs: 42130821.9.3001.5200
Record Dates: First submitted 2022-07-31; First posted 2022-10-10 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Respiratory Infection
Keywords: surface electromyography; EMGs; electromyography; coronavirus 2; SARS-CoV-2; Coronavirus; Intensive care unit; ICU; critically ill; Risk of orotracheal intubation; respiratory muscle fatigue; breathing muscles; EMG; COVID-19 Respiratory Infection
MeSH Terms: conditions — Coronavirus Infections; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Classification of oxygenation status stratification: Patients were classified into 3 groups with stratification of oxygenation status based on the relationship between blood oxygen saturation (SpO2) and fraction of inspired oxygen (FiO2) SpO2/FiO2, divided into three categories: normal (> 315), mild to moderate (314 - 235) and severe (< 234).

SUMMARY:
This research was characterized as a cross-sectional observational study, following the recommendations of the STROBE instrument. Therefore, it was conducted in the Intensive Care Unit of Otávio de Freitas Hospital (HOF) in Recife/PE, with patients over 18 years old who had a clinical diagnosis of COVID-19, using two methods of oxygen therapy (Nasal Oxygen Therapy) and (non-rebreather mask). Consequently, clinical evaluations were performed regarding the disease, severity of COVID-19, perception of respiratory effort, and electromyography of respiratory muscles.

1. Leading Question: How does the recruitment pattern of diaphragmatic and extradiaphragmatic muscles in patients with acute hypoxemia caused by COVID-19 behave when assessed through EMGs, considering the SpO2/FiO2 ratio as the analysis parameter?
2. Leading Question: Is there a relationship between the respiratory work estimated by electromyographic activity of diaphragmatic and extradiaphragmatic muscles in patients with acute hypoxemia due to COVID-19 and the parameters of respiratory frequency and levels of acute hypoxemia measured by the SpO2/FiO2 ratio?

The rationale for this study is that the COVID-19 pandemic has caused significant impacts on global public health due to the high volume of respiratory complications in the face of a limited supply of healthcare resources, consequently leading to high mortality. Complications are initially manifested by acute hypoxemia associated with COVID-19 infection, sometimes silent upon visual inspection or using less sensitive methods. This complicates the management of compensatory respiratory work for hypoxemia, even with oxygen therapy support. Respiratory muscle recruitment involves aspects of inspiratory effort and ventilatory mechanics. Recognizing the presence and recruitment pattern of muscles involved in a timely manner can contribute to the clinical management success rate of individuals affected by respiratory dysfunction associated with COVID-19, especially at different levels of acute hypoxemia. Surface electromyography is a non-invasive, low-risk tool compatible with the analysis of respiratory muscle recruitment patterns. However, there are no studies describing this pattern in COVID-19 patients, serving as a basis for personalized therapeutic strategies.

DETAILED DESCRIPTION:
1. GENERAL OBJECTIVE To analyze the clinical aspects of surface electromyography of respiratory muscles in COVID-19 patients under different levels of hypoxemia.
2. SPECIFIC OBJECTIVES To analyze the recruitment pattern of diaphragmatic and extradiaphragmatic muscles (sternocleidomastoid, scalene, and rectus abdominis) under different levels of acute hypoxemia in COVID-19 patients using the SpO2/FiO2 ratio as an analysis parameter and their relationships with clinical outcomes.
3. STUDY SITE AND PERIOD This study was conducted in the Intensive Care Unit in the Severe Acute Respiratory Syndrome (SARS) sector of Otávio de Freitas Hospital (HOF), located in the city of Recife, Pernambuco - Brazil.
4. SAMPLE The sample for this study consisted of spontaneously breathing patients admitted to the ICU diagnosed with COVID-19, who required low-flow oxygen therapy, using a nasal oxygen catheter or non-rebreathing mask.
5. CLINICAL EVALUATION At the beginning, a comprehensive clinical assessment was carried out which included the following parameters: name, assessment date, date of birth, address, telephone contact, age (years), sex (male/female), weight (kg), height (cm ), Body Mass Index (BMI - weight, kg / height², m²), Heart Rate (HR - bpm), Respiratory Rate (RR - rpm) assessed through chest expansibility (assessed visually for 1 minute), Systolic Blood Pressure (SBP - in mmHg), Diastolic Blood Pressure (DBP - in mmHg), Mean Arterial Pressure (MAP), Peripheral Oxygen Saturation (SpO2), method of administration in oxygen therapy, medications in use, other diagnoses, length of stay in the ICU , as well as outcomes of tracheal intubation and death were analyzed prospectively.
6. ASSESSMENT INSTRUMENTS Assessment of the severity of COVID-19 using the National Early Warning Score (NEWS2) and the Simplified Acute Physiological Score (SAPS3); Stratification of oxygenation status based on the relationship between blood oxygen saturation (SpO2) and the fraction of inspired oxygen (FiO2) SpO2/FiO2, divided into three categories: normal (> 315), mild to moderate (314 - 235) and severe (< 234); Assessment of the perception of respiratory effort using the modified Borg scale and assessment of respiratory work specific to COVID-19, which has been predicting the need for intubation; Evaluation of surface electromyography in the respiratory muscles, electrodes positioned in such a way that they aligned with the muscle fibers of the sternocleidomastoid, scalenes, diaphragm and rectus abdominis muscles.
7. RESULTS Independently of the severity of hypoxemia, the observed pattern of muscle recruitment remained similar between the groups, with higher RMS values for the extradiaphragmatic muscles (scalene and sternocleidomastoid), followed by the diaphragm and rectus abdominis muscles, respectively. When comparing the SpO2/FiO2 groups, significant differences were observed in the scalene and sternocleidomastoid muscles. The scalene muscles showed lower activation in mild-moderate and severe cases compared to the normal group, while the sternocleidomastoid also exhibited reduced activation in mild-moderate cases compared to the normal group. However, no differences were identified in the recruitment level of the diaphragm and rectus abdominis muscles among the SpO2/FiO2 groups.
8. ETHICAL ASPECTS This research project was approved by the Human Research Ethics Committee of the Federal University of Pernambuco (UFPE), where it complied with the postulates of the Declaration of Helsinki, following the terms recommended by the National Health Council (Resolution No. 466/ 2012) for research involving human subjects (approval number 4,560,383)

ELIGIBILITY:
Inclusion criteria:

* Both genders
* Age ≥ 18 years
* Confirmed diagnosis for COVID-19 considering its positivity through the RT-PCR test
* Patients who required low-flow oxygen therapy (nasal oxygen catheter or non-rebreathing mask)
* Hemodynamic stability (heart rate between 60 - 149 bpm, systolic blood pressure ≤149/89 mmHg or diastolic ≥ 90/60 mmHg at the time of collection)
* Body Mass Index ≤ 30 kg/m².

Exclusion criteria:

* Anxiety and psychomotor agitation
* Postural deformities (hyperlordosis, hyperkyphosis, lateral inclinations and antalgic postures)
* Patients with chronic lung disease or diaphragmatic disorders
* Undergoing surgical procedures on the spine
* Neurological diseases that affect myoelectric conduction
* Trauma or musculoskeletal injuries to the rib cage or respiratory muscles
* Use of tracheostomy tubes
* History of use of invasive mechanical ventilation during hospitalization (diagnosed and previously described in the electronic medical record)
* Those who were using sedatives and bronchodilators, as well as a reduction in SpO2 during signal acquisition at the time of collection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample of this study consisted of patients admitted to the ICU with spontaneous breathing diagnosed with COVID-19, who required low-flow oxygen therapy, using a nasal oxygen catheter or non-rebreathing mask.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Degree of dyspnea | 10 minutes
  Evaluate the degree of dyspnea using the modified Borg scale, which characterizes the respiratory fatigue reported by patients, characterizing the degree of dyspnea with scores from 0 to 10, where 0 is (no discomfort) and a maximum score of 10 (maximum discomfort).
Level of activation of respiratory muscles | 10 minutes
  As a way of analyzing the level of activation and fatigue of the respiratory muscles, surface electromyography (EMGS) was used in the respiratory muscles, analyzed using a surface electromyography, and the following muscles were evaluated: Sternocleidomastoid, scalene, diaphragm and rectus abdominis.

SECONDARY OUTCOMES:
Assessment of the perception of respiratory effort in COVID-19 | 10 minutes
  Assessing the perception of respiratory effort through a validated instrument to assess the work of breathing in COVID-19 (Apigo et al., 2020) has been predicting the need for orotracheal intubation, associating respiratory rate, nasal flaring and use of accessory respiratory muscles.

OTHER OUTCOMES:
Assessment of the severity of COVID -19 | 10 minutes
  To describe the severity of COVID -19 given by the National Early Warning Score (NEWS2) scale in three categories: Low risk (between 0 and 4 points), medium risk (between 5 and 6 points) and high risk greater (than 7 points).
  The assessment called Simplified Acute Physiological Score (SAPS3) aims to analyze the severity of the disease during the ICU stay, consisting of previous data on the health status, complications that led to hospitalization, information related to the physiological and laboratory tests during the ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Fernandes Ferreira da silva Júnior, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Physical Therapy Department, Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miralles R, Gamboa NA, Gutierrez MF, Santander H, Valenzuela S, Bull R, Fuentes AD, Cordova R. Effect of breathing type on electromyographic activity of respiratory muscles during tooth clenching at different decubitus positions. Cranio. 2019 Jan;37(1):28-34. doi: 10.1080/08869634.2018.1470274. Epub 2018 May 7. PMID 29730974
- [Result] Alonso JF, Mananas MA, Rojas M, Bruce EN. Coordination of respiratory muscles assessed by means of nonlinear forecasting of demodulated myographic signals. J Electromyogr Kinesiol. 2011 Dec;21(6):1064-73. doi: 10.1016/j.jelekin.2011.07.004. Epub 2011 Aug 6. PMID 21821430
- [Result] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Result] Apigo M, Schechtman J, Dhliwayo N, Al Tameemi M, Gazmuri RJ. Development of a work of breathing scale and monitoring need of intubation in COVID-19 pneumonia. Crit Care. 2020 Jul 31;24(1):477. doi: 10.1186/s13054-020-03176-y. No abstract available. PMID 32736637
- [Result] Beck J, Sinderby C, Lindstrom L, Grassino A. Diaphragm interference pattern EMG and compound muscle action potentials: effects of chest wall configuration. J Appl Physiol (1985). 1997 Feb;82(2):520-30. doi: 10.1152/jappl.1997.82.2.520. PMID 9049732
- [Result] Bissett B, Gosselink R, van Haren FMP. Respiratory Muscle Rehabilitation in Patients with Prolonged Mechanical Ventilation: A Targeted Approach. Crit Care. 2020 Mar 24;24(1):103. doi: 10.1186/s13054-020-2783-0. PMID 32204719
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Cabanes-Martinez L, Villadoniga M, Gonzalez-Rodriguez L, Araque L, Diaz-Cid A, Ruz-Caracuel I, Pian H, Sanchez-Alonso S, Fanjul S, Del Alamo M, Regidor I. Neuromuscular involvement in COVID-19 critically ill patients. Clin Neurophysiol. 2020 Dec;131(12):2809-2816. doi: 10.1016/j.clinph.2020.09.017. Epub 2020 Oct 15. PMID 33137571
- [Result] Caruso P, Albuquerque AL, Santana PV, Cardenas LZ, Ferreira JG, Prina E, Trevizan PF, Pereira MC, Iamonti V, Pletsch R, Macchione MC, Carvalho CR. Diagnostic methods to assess inspiratory and expiratory muscle strength. J Bras Pneumol. 2015 Mar-Apr;41(2):110-23. doi: 10.1590/S1806-37132015000004474. PMID 25972965
- [Result] Cecchini J, Schmidt M, Demoule A, Similowski T. Increased diaphragmatic contribution to inspiratory effort during neurally adjusted ventilatory assistance versus pressure support: an electromyographic study. Anesthesiology. 2014 Nov;121(5):1028-36. doi: 10.1097/ALN.0000000000000432. PMID 25208082
- [Result] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Result] Chiti L, Biondi G, Morelot-Panzini C, Raux M, Similowski T, Hug F. Scalene muscle activity during progressive inspiratory loading under pressure support ventilation in normal humans. Respir Physiol Neurobiol. 2008 Dec 31;164(3):441-8. doi: 10.1016/j.resp.2008.09.010. Epub 2008 Oct 4. PMID 18952011
- [Result] Palacios Cruz M, Santos E, Velazquez Cervantes MA, Leon Juarez M. COVID-19, a worldwide public health emergency. Rev Clin Esp. 2021 Jan;221(1):55-61. doi: 10.1016/j.rce.2020.03.001. Epub 2020 Mar 20. English, Spanish. PMID 32204922
- [Result] Da Gama AE, de Andrade Carvalho L, Feitosa LA, do Nascimento Junior JF, da Silva MG, Amorim CF, Aliverti A, Lambertz D, Rodrigues MA, de Andrade AD. Acute effects of incremental inspiratory loads on compartmental chest wall volume and predominant activity frequency of inspiratory muscle. J Electromyogr Kinesiol. 2013 Dec;23(6):1269-77. doi: 10.1016/j.jelekin.2013.07.014. Epub 2013 Aug 11. PMID 24035013
- [Result] Daimon S, Yamaguchi K. Changes in respiratory activity induced by mastication during oral breathing in humans. J Appl Physiol (1985). 2014 Jun 1;116(11):1365-70. doi: 10.1152/japplphysiol.01236.2013. Epub 2014 Apr 17. PMID 24744386
- [Result] Dionne A, Parkes A, Engler B, Watson BV, Nicolle MW. Determination of the best electrode position for recording of the diaphragm compound muscle action potential. Muscle Nerve. 2009 Jul;40(1):37-41. doi: 10.1002/mus.21290. PMID 19533636
- [Result] Dos Reis IMM, Ohara DG, Januario LB, Basso-Vanelli RP, Oliveira AB, Jamami M. Surface electromyography in inspiratory muscles in adults and elderly individuals: A systematic review. J Electromyogr Kinesiol. 2019 Feb;44:139-155. doi: 10.1016/j.jelekin.2019.01.002. Epub 2019 Jan 11. PMID 30658230
- [Result] Drake JD, Callaghan JP. Elimination of electrocardiogram contamination from electromyogram signals: An evaluation of currently used removal techniques. J Electromyogr Kinesiol. 2006 Apr;16(2):175-87. doi: 10.1016/j.jelekin.2005.07.003. Epub 2005 Aug 31. PMID 16139521
- [Result] Dres M, Schmidt M, Ferre A, Mayaux J, Similowski T, Demoule A. Diaphragm electromyographic activity as a predictor of weaning failure. Intensive Care Med. 2012 Dec;38(12):2017-25. doi: 10.1007/s00134-012-2700-3. Epub 2012 Sep 26. PMID 23011532
- [Result] Duiverman ML, de Boer EW, van Eykern LA, de Greef MH, Jansen DF, Wempe JB, Kerstjens HA, Wijkstra PJ. Respiratory muscle activity and dyspnea during exercise in chronic obstructive pulmonary disease. Respir Physiol Neurobiol. 2009 Jun 30;167(2):195-200. doi: 10.1016/j.resp.2009.04.018. Epub 2009 May 3. PMID 19406254
- [Result] Falla D, Dall'Alba P, Rainoldi A, Merletti R, Jull G. Location of innervation zones of sternocleidomastoid and scalene muscles--a basis for clinical and research electromyography applications. Clin Neurophysiol. 2002 Jan;113(1):57-63. doi: 10.1016/s1388-2457(01)00708-8. PMID 11801425
- [Result] Gallego J, Perez de la Sota A, Vardon G, Jaeger-Denavit O. Electromyographic feedback for learning to activate thoracic inspiratory muscles. Am J Phys Med Rehabil. 1991 Aug;70(4):186-90. doi: 10.1097/00002060-199108000-00005. PMID 1878176
- [Result] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Result] Hutten GJ, van Thuijl HF, van Bellegem AC, van Eykern LA, van Aalderen WM. A literature review of the methodology of EMG recordings of the diaphragm. J Electromyogr Kinesiol. 2010 Apr;20(2):185-90. doi: 10.1016/j.jelekin.2009.02.008. Epub 2009 May 6. PMID 19423360
- [Result] Segizbaeva MO, Aleksandrova NP. [Inspiratory muscle resistance to fatigue during exercise and simulated airway obstruction]. Fiziol Cheloveka. 2014 Nov-Dec;40(6):114-22. Russian. PMID 25711114
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. Addendum: A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Dec;588(7836):E6. doi: 10.1038/s41586-020-2951-z. No abstract available. PMID 33199918